IRB Protocol Number: 2019H0092
IRB Approval date: XXX
Version: 07/19/21

## The Ohio State University Consent to Participate in Research

Online Implementation Survey

**Determinants of Implementation Success Coordinating** 

Study Title: Ventilator, Early Ambulation and Rehabilitation Efforts in the

ICU (DISCOVER-ICU)

**Researcher:** Lorraine Mion, PhD, RN, FAAN

**Sponsor:** National Heart, Lung, and Blood Institute (NIH)

3 4

1

This is a consent form for research participation. It contains important information about this study and what to expect if you decide to participate.

5 6 7

Your participation is voluntary.

8 9

Please consider the information carefully. Feel free to ask questions before making your decision whether or not to participate.

10 11 12

13

14

15

16 17

18 19 **Purpose:** The purpose of the DISCOVER-ICU study is to develop multilevel implementation strategies to enhance sustainable uptake of the ABCDEF bundle into routine clinical practice. This survey provides the name and definition of variable actions/strategies used to increase adoption of evidence-based intensive care unit (ICU) practices. We are interested in learning what actions/strategies your ICU team used to facilitate adoption of the ABCDEF bundle during the course of time you spent participating in the Society of Critical Care Medicine's ICU Liberation Collaborative that began on August 1<sup>st</sup>, 2015 and concluded on April 30<sup>th</sup>, 2017. We are also interested in discovering whether your team found these actions/strategies helpful, acceptable, feasible, and costly.

202122

23

24

25

**Procedures/Tasks:** We ask that you engage colleagues from various disciplines (e.g., nursing, medicine, pharmacy, respiratory/physical/occupational therapy) who worked in your unit during the ICU Liberation Collaborative in completion of the survey. There is no set approach in garnering your team's input. We encourage you to do what is best for you and your ICU team. You may choose to:

262728

29

3031

32

33

34

- 1) Conduct a meeting specifically focused on completing the online survey. During this team meeting, the online survey could be accessed, questions discussed, and responses entered simultaneously. We recommend this approach as it is likely to be the most comprehensive and least time consuming.
- 2) Print a hardcopy of the survey to discuss and complete during a regularly scheduled or small group team meeting. Once the survey is complete, one team member would then enter the site data into the online survey.

IRB Protocol Number: 2019H0092
IRB Approval date: XXX
Version: 07/19/21

3) Print hardcopies of the survey and ask each team member to complete it individually. Once responses are received, one team member would then resolve any conflicting answers and enter the site data into the online survey.

4) Distribute a word or PDF version of the survey via email communication to team members. Completed surveys could then be given to one team member who would then would resolve any conflicting answers and enter the site data into the online survey.

There may be some disagreements among professionals on various aspects of the survey. Because only one survey may be submitted per site, we ask you complete it as well as you can and as closely aligned with the team's consensus as possible. If necessary, we suggest the team member who played the most active role in ABCDEF bundle implementation efforts resolves any disagreements.

 **Duration:** Because we are requesting the engagement of multiple stakeholders, we anticipate that the time necessary to complete the survey may vary by site. We estimate it will take approximately 20 minutes for an individual to complete the survey and approximately 40-50 minutes to complete the survey if discussed during a team meeting.

You may leave the study at any time. If you decide to stop participating in the study, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. Your decision will not affect your future relationship with The Ohio State University.

**Risks and Benefits:** There are no known physical or psychologic risks to being in the study. You may skip any survey questions you do not wish to answer.

You will not receive any benefit from study participation, but your opinions and experiences may contribute to a better understanding of what strategies are most beneficial in terms of increasing ABCDEF bundle adoption.

**Confidentiality:** We will work to make sure that no one sees your online responses without approval. But, because we are using the Internet, there is a chance that someone could access your online responses without permission. In some cases, this information could be used to identify you.

Your data will be protected with a code to reduce the risk that other people can view the responses.

 Also, there may be circumstances where this information must be released. For example, personal information regarding your participation in this study may be disclosed if required by state law. Also, your records may be reviewed by the following groups (as applicable to the research):

IRB Protocol Number: 2019H0092
IRB Approval date: XXX

Version: 07/19/21

• Office for Human Research Protections or other federal, state, or international regulatory agencies;

- The Ohio State University Institutional Review Board or Office of Responsible Research Practices:
- The sponsor, if any, or agency (including the Food and Drug Administration for FDA-regulated research) supporting the study.

Future Research: Your de-identified information may be used or shared with other researchers without your additional informed consent.

**Incentives:** Each team member who participates in completing the survey, maximum of four team members per site, will receive a \$25 Amazon gift card. In addition, the person responsible for entering the site data into REDCap will receive an additional \$25 Amazon gift card. Reimbursement will occur once all of the survey data is entered into REDCap.

By law, payments to participants are considered taxable income.

**Participant Rights:** You may refuse to participate in this study without penalty or loss of benefits to which you are otherwise entitled. If you are a student or employee at Ohio State, your decision will not affect your grades or employment status.

If you choose to participate in the study, you may discontinue participation at any time without penalty or loss of benefits. By agreeing to participate, you do not give up any personal legal rights you may have as a participant in this study.

An Institutional Review Board responsible for human subjects research at The Ohio State University reviewed this research project and found it to be acceptable, according to applicable state and federal regulations and University policies designed to protect the rights and welfare of participants in research.

**Contacts and Questions:** For questions, concerns, or complaints about the study, or you feel you have been harmed as a result of study participation, you may contact Dr. Lorraine Mion via email at mion.3@osu.edu or by telephone at 614-688-3734.

## **Providing consent**

I have read (or someone has read to me) this page and I am aware that I am being asked to participate in a research study. I have had the opportunity to ask questions and have had them answered to my satisfaction. I voluntarily agree to participate in this study. I am not giving up any legal rights by agreeing to participate.

CONSENT IRB Protocol Number: 2019H0092
Biomedical/Cancer IRB Approval date: XXX
Version: 07/19/21

To print or save a copy of this page, select the print button on your web browser.

122123

Please click the button below to proceed and participate in this study. If you do not wish to participate, please close out your browser window.

124 125 126